CLINICAL TRIAL: NCT06591078
Title: Clinical Efficacy Evaluation and Mechanism Study of Potential Advantageous Diseases of Acupuncture - Evaluation of Clinical Efficacy of Acupuncture in Improving Immune Response in Patients With Cervical Cancer
Brief Title: Evaluation of Clinical Efficacy of Acupuncture in Improving Immune Response in Patients With Cervical Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ying Zhang (Other)
Collaborators: Peking Union Medical College Hospital (Other); Beijing Obstetrics and Gynecology Hospital (Other); Peking University Cancer Hospital & Institute (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Sichuan Cancer Hospital and Research Institute (Other); Shanghai University of Traditional Chinese Medicine (Other); Hunan Cancer Hospital (Other); Chongqing University Cancer Hospital (Other)
Responsible Party: Sponsor-Investigator, Ying Zhang, Director, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Organization: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HLCMMHPP2023089-08
Record Dates: First submitted 2024-06-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cervical Cancer
Keywords: Acupuncture; immunotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): 1.Carrilizumab for injection; 200mg; Q14d; 2.Apatinib; 250mg Qd or Bid or chemotherapy; 3.electropuncture; 4/Q28d.
  Use up to 2 years/ patient disease progression(about 1 year)/ unacceptable toxic effects, use of prohibited therapies (such as antitumor therapy other than chemotherapy and beva or non-palliative radiotherapy)/ investigator's decision to discontinue the regimen/ or patient's withdrawal of consent treatment may be discontinued. If a patient with a confirmed complete response has received at least eight cycles of immunotherapy, including at least two cycles beyond a complete response, treatment will be discontinued.
  Interventions: Other: electropuncture
- control group (No Intervention): 1.Carrilizumab for injection; 200mg; Q14d; 2.Apatinib; 250mg Qd or Bid or chemotherapy; Use up to 2 years/ patient disease progression(about 1 year)/ unacceptable toxic effects, use of prohibited therapies (such as antitumor therapy other than chemotherapy and beva or non-palliative radiotherapy)/ investigator's decision to discontinue the regimen/ or patient's withdrawal of consent treatment may be discontinued. If a patient with a confirmed complete response has received at least eight cycles of immunotherapy, including at least two cycles beyond a complete response, treatment will be discontinued.

INTERVENTIONS:
Other: electropuncture — The needle was retained for 30 minutes. During the retention period, the needle was lifted and twisted for 3 times with even small amplitude every 10 minutes, and the complement method was performed for 3 times. No manipulation before the needle, cotton ball press directly out of the needle.
  ④ Frequency, course and time: Start at the same time as immunotherapy, and complete 1-2 times of electroacupuncture treatment per week; Electroacupuncture was performed 4 times per 28 days. The number of electroacupuncture treatment cycles and the number of immunotherapy courses should be consistent.
  Arms: experimental group

SUMMARY:
In a prospective, multicenter, randomized, controlled study, patients with metastatic, recurrent, or persistent cervical cancer who were ineligible for surgery and/or radiotherapy were randomly assigned in a 1:1 ratio to either an experimental group or a control group." The control group was treated with apatinib combined with callizumab/callizumab combined with chemotherapy, and the experimental group was treated with electroacupuncture on the basis of the treatment. Anti-tumor efficacy, immune function efficacy, quality of life and safety were used as the outcome indicators.

DETAILED DESCRIPTION:
1. Study Design Types:

   This was a prospective, multicenter, randomized controlled clinical study.
2. Random method:

   This study used central randomization method. A total of 90 patients with recurrent/metastatic cervical cancer were enrolled and divided into 8 research centers. Patients were divided into control group (group A) and experimental group (group B) according to the pathological type, PD-L1 expression level, immunotherapy combined with targeted therapy/immunotherapy combined with chemotherapy as stratification factors at each research center. The block length was 6, and the allocation ratio was 1∶1.
3. Control methods:

   This trial included a control group and an experimental group. The intervention measures of the experimental group included acupuncture + immunotherapy + targeted therapy/acupuncture + immunotherapy + chemotherapy. The intervention measures of the control group were immunotherapy + targeted therapy/immunotherapy + chemotherapy.
4. Sample size calculation:

This study intends to conduct preliminary exploratory research and use small samples for clinical observation. The sample size of each group of exploratory research should be more than 30 according to literature. This exploratory study intends to include 90 patients to be allocated to the experimental group and the control group

ELIGIBILITY:
Inclusion Criteria:

1. Patients with metastatic, recurrent or persistent cervical cancer including squamous cell carcinoma, adenosquamous cell carcinoma, that is not suitable for surgery and/or radiation therapy;
2. Age 18-70 years old;
3. Have at least one measurable lesion according to RECIST 1.1; Note: Measurable lesions are defined as those that can be accurately measured in at least one dimension (the longest diameter recorded by computed tomography (CT) scanning, magnetic resonance imaging (MRI) is ≥10mm; Lymph nodes must be ≥15mm on the short axis. Tumors within the previously irradiated area will be designated as "off-target" lesions unless progress is recorded at least 90 days after completion of radiation therapy or a biopsy is performed to confirm persistence.
4. The ECOG score is 0 or 1;
5. Life expectancy exceeds 3 months;
6. The patient's important organs function normally, as follows:

   Absolute neutrophil count (ANC) ≥1.5×10^9/L; Platelet count ≥80×10^9/L; Hemoglobin ≥90g/L;

   ④ Total bilirubin ≤1.5× upper limit of normal (ULN);

   ⑤ Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN; Note: In patients with liver metastasis, AST and ALT levels were ≤5 ×ULN;

   ⑥ Creatinine ≤1.5×ULN or creatinine clearance ≥60 ml/min (Cockcroft-Gault formula);

   ⑦ Baseline albumin ≥28g/L;
7. Thyroid stimulating hormone (TSH) level ≤1×ULN; Note: Patients with free triiodothyronine [FT3] or free thyroxine [FT4] levels ≤1× ULN may be included.
8. Patients can sign written informed consent.

Exclusion Criteria:

1. histopathological diagnosis of squamous cell carcinoma, adenosquamous carcinoma, or tumors other than adenocarcinoma;
2. have participated in another clinical trial, or completed another clinical trial within 4 weeks;
3. previous use of immune checkpoint inhibitors, including but not limited to other anti-PD-1 and anti-PD-L1 antibodies;
4. a known history of allergy to any component of carrilizumab preparations or other monoclonal antibodies;
5. Immunosuppressive drugs are currently required; Note: Prednisone > 10 mg/d or equivalent dose is prohibited within 2 weeks prior to administration of the study drug.
6. Patients with any active autoimmune disease or history of autoimmune disease, including but not limited to the following: hepatitis, pneumonia, uveitis, colitis (inflammatory bowel disease), pituitaritis, vasculitis, nephritis, hyperthyroidism and hypothyroidism, asthma patients requiring intermittent use of bronchodilators or other medical interventions; Note: Excluding vitiligo, resolved childhood asthma/atopic subjects.
7. Clinically significant cardiovascular disease, including but not limited to congestive heart failure (NYHA level > 2), unstable or severe angina, severe acute myocardial infarction within 1 year prior to enrollment, supraventricular or ventricular arrhythmias requiring medical intervention, or QT interval ≥470 milliseconds (women);
8. Arterial thrombosis or venous thrombosis occurs within 6 months; Hypertension medications do not adequately control hypertension (systolic blood pressure ≥140 mm Hg and/or diastolic blood pressure ≥90 mm Hg);

(10) proteinuria ≥ (++) or 24-hour urinary protein total > 1.0g; (11) Abnormal coagulation (INR > 2.0, PT > 16s), bleeding tendency or receiving thrombolytic or anticoagulant therapy; (12) has not recovered from an adverse event (other than hair loss) from prior administration (i.e. ≤ Grade 1 or baseline); (13) Known active central nervous system metastases; (14) Patients with prior invasive malignancy and any evidence of disease within the past 5 years; Note: Exceptions are basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or cervical cancer in situ that has received potentially curative treatment.

(15) Have an active infection that requires systemic treatment; (16) A history of immunodeficiency, including seropositivity for human immunodeficiency virus (HIV) or other acquired or congenital immunodeficiency diseases; Hepatitis B virus (HBV) > 2000 IU/ml or DNA≥1×10^4/ml; Or hepatitis C virus (HCV) RNA ≥1×10^3/ml); (18) Received live vaccine within 4 weeks before the first trial treatment; Note: Inactivated virus vaccines against seasonal influenza are allowed. (19) Patients with suspected intestinal obstruction or risk of vagino-rectal fistula or vagino-vesical fistula; (20) Any other medical, mental, or social condition that the investigator believes may interfere with the subject's rights, safety, welfare, or ability to sign informed consent, cooperate, and participate in the study, or with the interpretation of the results.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
objective remission rate | The patients were evaluated every 8 weeks ±2 weeks from the beginning of treatment until 40 weeks, and then every 12 weeks ±2 weeks until the end of treatment.
  ORR refers to the proportion of patients whose tumor volume has shrunk to a predetermined value and can maintain the minimum time required. Cases with complete response (CR) and partial response (PR) were included.

SECONDARY OUTCOMES:
progression free survival | The patients were evaluated every 8 weeks ±2 weeks from the beginning of treatment until 40 weeks, and then every 12 weeks ±2 weeks until the end of treatment.
  ORR refers to the proportion of patients whose tumor volume has shrunk to a predetermined value and can maintain the minimum time required. Cases with complete response (CR) and partial response (PR) were included.
overall survival | The patients were followed up until death or at least 2 years
  From randomization to the time of death from any cause.
disease control rate | The patients were evaluated every 8 weeks ±2 weeks from the beginning of treatment until 40 weeks, and then every 12 weeks ±2 weeks until the end of treatment.
  DCR refers to the proportion of patients whose tumor volume has shrunk or stabilized to a predetermined value and can maintain the minimum time required. Cases with complete response (CR), partial response (PR), and stable disease (SD) were included
Tumor marker | The patients were evaluated every 8 weeks ±2 weeks from the beginning of treatment until 40 weeks, and then every 12 weeks ±2 weeks until the end of treatment.
  Tumor marker level of CA 125 and SCC.
Quality of life improvement | The patients were evaluated every 8 weeks ±2 weeks from the beginning of treatment until 40 weeks, and then every 12 weeks ±2 weeks until the end of treatment.
  Use scale to evaluated the quality of life of patients.
Adverse events associated with immunotherapy and targeted therapy and their severity | The patients were evaluated every 8 weeks ±2 weeks from the beginning of treatment until 40 weeks, and then every 12 weeks ±2 weeks until the end of treatment.
  NCI CTCAE V5.0 evaluation criteria for adverse events, including but not limited to skin reactions, pneumonia, colitis, nephritis, endocrine diseases, etc
Security Index | he patients were evaluated every 8 weeks ±2 weeks from the beginning of treatment until 40 weeks, and then every 12 weeks ±2 weeks until the end of treatment.
  Blood, urine, stool routine, liver function (ALT, AST), kidney function (Cr, BUN) examination.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Zhang, phd, Study Director — Guang 'anmen Hospital, China Academy of Chinese Medical Sciences

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT06591078/Prot_SAP_000.pdf
  • Informed Consent Form (2024-07-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT06591078/ICF_001.pdf